CLINICAL TRIAL: NCT01844557
Title: Testing Accountability in Patient Adherence
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2013-0195; 5R01DE019141-03 (NIH)
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Head And Neck Cancer
Keywords: Head And Neck Cancer; Nasopharyngeal cancer; Oropharyngeal cancer; Hypopharyngeal cancer; Laryngeal cancer; Primary cancer with cervical metastases; Swallowing exercises; Videotape; Videocamera; M.D. Anderson Symptom Inventory; Questionnaires; Surveys
MeSH Terms: conditions — Head and Neck Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group 1(High Accountability-Human Monitoring): Participants randomly assigned to receive one of three sets of instructions before starting. Instructions for three swallowing exercises as well as an introductory script explaining the purpose of the exercises will be videotaped and shown to participants. Participants perform 3 swallowing exercises while researcher leaves the room. At the end of the testing period, researcher will come back into the room and record the number on participant's tracking device. Participant to tell whether they did as many repetitions as possible and if not, why they were not able to do as many as possible. This portion of the experiment will be videotaped. Participants complete an M.D. Anderson Symptom Inventory for Head and Neck Cancer Patients before procedure as well as a brief 3-page post-session questionnaire.
  Interventions: Other: Swallowing Exercises; Behavioral: Symptom Inventory; Behavioral: Questionnaires
- Group 2(Low Accountability-Human Monitoring): Participants randomly assigned to receive one of three sets of instructions before starting. Instructions for three swallowing exercises as well as an introductory script explaining the purpose of the exercises will be videotaped and shown to participants. Participants perform 3 swallowing exercises while researcher leaves the room. At the end of the testing period, researcher will come back into the room and record the number on participant's tracking device. Participants complete an M.D. Anderson Symptom Inventory for Head and Neck Cancer Patients before procedure as well as a brief 3-page post-session questionnaire.
  Interventions: Other: Swallowing Exercises; Behavioral: Symptom Inventory; Behavioral: Questionnaires
- Group 3(Low Accountability-Technological Monitoring): Participants randomly assigned to receive one of three sets of instructions before starting. Instructions for three swallowing exercises as well as an introductory script explaining the purpose of the exercises will be videotaped and shown to participants. Participants perform 3 swallowing exercises while researcher leaves the room. At the end of the testing period, researcher will come back into the room and record the number on participant's tracking device. The videocamera will tape participant's session so evaluation can be made as to exercise accuracy. Participants complete an M.D. Anderson Symptom Inventory for Head and Neck Cancer Patients before procedure as well as a brief 3-page post-session questionnaire.
  Interventions: Other: Swallowing Exercises; Behavioral: Symptom Inventory; Behavioral: Questionnaires

INTERVENTIONS:
Other: Swallowing Exercises — Participants perform 3 swallowing exercises.
Behavioral: Symptom Inventory — Participants complete an M.D. Anderson Symptom Inventory for Head and Neck Cancer Patients before swallowing exercise procedure.
Behavioral: Questionnaires — Participants fill out 3 questionnaires after swallowing exercises. The questionnaires will take about 10 minutes to complete.
  Other Names: Surveys

SUMMARY:
The goal of this research study is to look for factors that influence whether or not head and neck cancer patients follow the swallowing exercises that they are asked to perform while receiving radiation treatment.

DETAILED DESCRIPTION:
Head and neck cancer patients who receive radiation are at risk for permanent swallowing disorders. Because of these potential problems, swallowing exercises are an important part of recovery. Researchers want to learn what factors affect how well patients follow the swallowing schedule they are given, and what can be done to make it consistent.

If you agree to take part in this study, you will have the following procedures performed.

Videotaped Swallowing Exercise:

Researchers will ask you to perform 3 swallowing exercises while being recorded by a video camera. The length of the taping session will be 3 minutes. Afterward, you will fill out 3 questionnaires. The questionnaires will take about 10 minutes to complete.

Length of Study:

You will be asked to come in 1 time for this study.

For the next 2 years, information may be collected from your medical record. This information will include the cancer stage, if the disease has gotten worse, any treatment you receive, and any side effects you experience. This information will help researchers learn how certain treatments affect patients and their risk for future disease.

This is an investigational study.

Up to 225 patient will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Are dispositioned to receive radiation with curative intent for nasopharyngeal, oropharyngeal, hypopharyngeal, laryngeal, or an unknown primary cancer with cervical metastases.
2. Are stage II-IVB for oropharyngeal and laryngeal
3. Are stage I-IVB for hypopharyngeal and nasopharyngeal
4. At least 18 years of age
5. Speak and read English
6. Oriented to time, person, and place
7. Have a Zubrod performance status of 0 to 2

Exclusion Criteria:

1. Have other cancer diagnoses, except non-melanoma skin cancer
2. Had treatment for previous H & N cancer or radiation to the head and neck
3. Have a history of previous head and neck surgery (excluding biopsy and/or tonsillectomy and/or tracheotomy)
4. Have a current oropharyngeal dysphagia unrelated to cancer diagnosis (e.g., dysphagia due to underlying neurogenic disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Head and neck cancer patients receiving radiation therapy at MDACC clinics.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to Swallowing Exercises | 1 day
  Purpose of experiment is to determine whether an accountability manipulation and whether human vs technological monitoring result in higher patient adherence. Main outcome measure is perseverance of effort which will be number of repetitions within one minute interval for each exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen H. Shinn, PHD, MS, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org